CLINICAL TRIAL: NCT06407323
Title: Pediatric Rehabilitation for Children With Cerebral Palsy Through Personalized Vibration Therapy Powered By Artificial Intelligence: An Innovative Approach to Reduce Spasticity and Improved Motor Function and Quality Of Life
Brief Title: Pediatric Rehabilitation for Children With Cerebral Palsy Through PVT Using AI to Reduce Spasticity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/704
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized vibration therapy powered by AI (Experimental)
  Interventions: Diagnostic Test: Personalized vibration therapy powered by AI
- physical therapy treatment (Other)
  Interventions: Other: Physical therapy treatment

INTERVENTIONS:
Diagnostic Test: Personalized vibration therapy powered by AI — A target frequency of either 20 Hz or 25 Hz, and amplitude 2-4 mm The whole treatment session will be around 20 minutes along with hot pack as a baseline treatment, consisted of 6 sessions per week for total 8 weeks of duration
  Arms: Personalized vibration therapy powered by AI
Other: Physical therapy treatment — A selected physical therapy treatment program for spastic diplegic CP.
  Arms: physical therapy treatment

SUMMARY:
The study foucs on pediatric rehabilitation for children with cerebral palsy through personalized vibration therapy powered by artificial intelligence.

DETAILED DESCRIPTION:
Innovative approach to reduce spasticity, improved motor function, quality of life. Vibration therapy reduces spasticity by activating the body's natural stretch reflex, which in turn triggers muscular contractions. Furthermore, it has been proposed that the primary ends of the muscle spindle Ia afferent are stimulated by muscular vibration. This leads to the excitation of alpha motor neurons, subsequent contractions of motor units, ultimately producing a tonic muscle contraction. This study will modify vibration therapy by introducing Artificial intelligence to rehabilitate the patients suffering from spastic CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed spastic CP as per neurologist report, GMFCS level I-III
* Ability to safely withstand intensity of vibrating device.
* have no planned surgery within 5 months before/after entering the study

Exclusion Criteria:

* A bone fracture within 12 weeks of enrollment.
* History of using anabolic agents, glucocorticoids (excluding inhaled), or growth hormone (regardless of dose) for at least 1 month, within the 3 months prior to enrollment.
* History of botulinum toxin injection into the lower limb(s) within the 3 months before enrollment.
* History of an illness or findings on physical examination that might prevent the child from completing the study (e.g., acute thrombosis, tendinitis).

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 12 Months
  It is used to assess spasticity of neurological disorder patients. For scores on the Modified Ashworth Scale, there was satisfactory inter- and intra-rater agreement. The results of the Modified Ashworth Scale showed more reliability in measuring the upper extremities than the lower. The inter-rater reliability of the ratings for the lower and upper extremities was statistically correlated with a number of study parameters
Quality of life-child Questionnaire | 12 months
  The first health condition-specific questionnaire created specifically to measure quality of life (QOL) in children with cerebral palsy (CP) is the Cerebral Palsy Quality of Life for Children (CP QOL-Child). For primary carers, intra-class correlation values varied from.88 to.97, while for children, they were between.91 and.98. The assessment of children with cerebral palsy (CP) using the Turkish version of the CP QOL questionnaire was found to be a valid and dependable method. b)Gross Motor Function Classification System There was 0.84 interrater reliability. The GMFCS level and motor development tests had a stronger correlation than the GMFCS level and non-motor development tests.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Johar pain relief center, Lahore, Punjab Province
  - Ali Fatima hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No